CLINICAL TRIAL: NCT05077527
Title: Axicabtagene Ciloleucel in Relapsed or Refractory HIV-Associated Aggressive B-Cell Non-Hodgkin Lymphoma
Brief Title: Immune Cell Therapy (CAR-T) for the Treatment of Patients With HIV and B-Cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-112; NCI-2021-02771 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-112 (Other: AIDS Malignancy Consortium); AMC-112 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: AIDS-Related Diffuse Large B-cell Lymphoma; AIDS-Related Non-Hodgkin Lymphoma; HIV Infection; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Grade 3b Follicular Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Transformed B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Grade 3b Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Transformed B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — HIV Infections; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — axicabtagene ciloleucel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (conditioning, axicabtagene ciloleucel) (Experimental): Patients receive fludarabine IV over 30 minutes and cyclophosphamide IV over 1 hour on days -5, -4, and -3. Patients then receive axicabtagene ciloleucel IV over 30 minutes on day 0.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — Given IV
  Other Names: KTE C19; KTE-C19; KTE-C19 CAR; Yescarta
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa

SUMMARY:
This phase I trial evaluates the side effects and usefulness of axicabtagene clioleucel (a CAR-T therapy) and find out what effect, if any, it has on treating patients with HIV-associated aggressive B-cell non-Hodgkin lymphoma that has come back (relapsed) or not responded to treatment (refractory). T cells are infection fighting blood cells that can kill tumor cells. Axicabtagene ciloleucel consists of genetically modified T cells, modified to recognize CD-19, a protein on the surface of cancer cells. These CD-19-specific T cells may help the body's immune system identify and kill CD-19-positive B-cell non-Hodgkin lymphoma cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate safety and feasibility of axicabtagene ciloleucel for relapsed/refractory (R/R) human immunodeficiency virus (HIV)-associated aggressive B-cell non-Hodgkin lymphoma (B-NHL) in participants with well-controlled HIV.

SECONDARY OBJECTIVES:

I. To estimate efficacy of axicabtagene ciloleucel in HIV-associated B-NHL as measured by complete response rate, event-free survival, and duration of response.

II. To assess the relationship between T-cell subset profile and clinical response in R/R HIV-associated B-NHL treated with axicabtagene ciloleucel.

EXPLORATORY OBJECTIVES:

I. To assess the relationship between immune-mediated response and clinical response and toxicity in HIV-associated B-NHL treated with axicabtagene ciloleucel.

II. To define burden of HIV integration in the final chimeric antigen receptor (CAR) T-cell product versus the pheresis product through quantitative polymerase chain reaction (PCR).

OUTLINE:

Patients receive fludarabine intravenously (IV) over 30 minutes and cyclophosphamide IV over 1 hour on days -5, -4, and -3. Patients then receive axicabtagene ciloleucel IV over 30 minutes on day 0.

After completion of study treatment, patients are followed up once weekly for month 1, once a month for months 2-6, and then at 9, 12, 15, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant with age >= 18 years at the time of consent. Because no dosing or adverse event data are currently available on the use of axicabtagene ciloleucel in participants < 18 years of age, children are excluded from this study
* Participant is able to understand and willing to sign a written informed consent document before any study procedures
* Participant must have R/R aggressive B-cell NHL of the following histologies:

  * Diffuse large B-cell lymphoma (DLBCL, including transformed from indolent histology)
  * High-grade B-cell lymphoma
  * Primary mediastinal B-cell lymphoma
  * Follicular lymphoma, grade 3B
* Participant must have been treated with an anthracycline and rituximab (or other CD20-targeted agent) and have R/R disease after at least 2 lines of therapy

  * At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic cancer therapy at the time the subject provides consent
* Evaluable disease as either:

  * Positron emission tomography (PET)-positive disease according to the "Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification", or
  * Bone marrow involvement assessed by bone marrow biopsy
* Eastern Cooperative Oncology Group ECOG performance status =< 1 (Karnofsky >= 60%)
* Serum creatinine =< 1.5 x age-adjusted upper limit of normal (ULN) OR calculated creatinine clearance (Cockcroft and Gault) > 30 mL/min/1.73 m^2 (within 4 weeks before enrollment)
* Alanine aminotransferase (ALT) =< 5 x ULN and total bilirubin < 2.0 mg/dL (or < 3.0 mg/dL for subjects with Gilbert's syndrome or lymphomatous infiltration of the liver or if taking atazanavir or indinavir (within 4 weeks before enrollment)
* Adequate pulmonary function, defined as =< Common Terminology Criteria for Adverse Events (CTCAE) grade 1 dyspnea and oxygen saturation (SaO2) >= 92% on room air (within 4 weeks before enrollment)
* Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) >= 40% as assessed by echocardiogram or multiple uptake gated acquisition (MUGA) scan performed within 1 month of determination of eligibility
* Absolute neutrophil count: >= 1,000/mm^3 (within 4 weeks before enrollment)
* Platelets: >= 75,000/mm^3 (within 4 weeks before enrollment)
* Total bilirubin: =< 1.5 x institutional upper limit of normal (ULN) (3.0 x ULN for patients with Gilbert syndrome) If, however, the elevated bilirubin is felt to be secondary to antiretroviral therapy, the total bilirubin must be =< 3.5 mg/dL, provided that the direct bilirubin is normal and the aspartate aminotransferase (AST) and ALT =< 3 x the upper limit of normal (within 4 weeks before enrollment)
* Adequate vascular access for leukapheresis procedure and for administration of the cellular product (either peripheral line or leukapheresis catheter)
* Participants who have received previous CD19-targeted therapy must have CD19-positive lymphoma confirmed on a biopsy since completing the prior CD19-targeted therapy
* The effects of axicabtagene ciloleucel on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) before study entry, for the duration of study participation, and 12 months after the last dose of axicabtagene ciloleucel. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Men who have partners of childbearing potential must agree to use an effective barrier contraceptive method before study entry, for the duration of study participation, and for 1 year after the last dose of axicabtagene ciloleucel
* Documentation of HIV-1 infection by means of any one of the following:

  * Documentation of HIV diagnosis in the medical record by a licensed health care investigator;
  * Documentation of receipt of antiretroviral therapy (ART) (at least two different medications that do not constitute a prescription for pre-exposure prophylaxis [PrEP]) by a licensed health care investigator. Documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name;
  * HIV-1 ribonucleic acid (RNA) detection by a licensed HIV-1 RNA assay demonstrating >1000 RNA copies/mL;

    * Any federally approved, licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay. NOTE: A "licensed" assay refers to a U.S. Food and Drug Administration (FDA)-approved assay, which is required for all Investigational New Drug (IND) studies
* HIV viral load below 50 copies/mL by FDA-approved assays within 4 weeks prior to registration
* A CD4 cell count must be obtained within 4 weeks before enrollment at any U.S. laboratory that has a clinical laboratory improvement amendments (CLIA) certification or its equivalent. Twenty participants will be studied with a goal to enroll a minimum of 6 participants with a CD4 <100 cells/uL
* Participants who have hepatitis C (reactive anti-HCV antibody) and hepatitis B (HBsAg positive and/or anti-HBc-Total positive), may be enrolled, provided total bilirubin is =< 1.5 x institutional upper limit of normal (ULN), AST (serum glutamic oxaloacetic transaminase [SGOT]) and ALT (serum glutamic pyruvic transaminase [SGPT]) must be =< 3 X institutional upper limit of normal, and HBV deoxyribonucleic acid (DNA) <100 IU/mL (if hepatitis B positive) within 4 weeks before enrollment. There must be no evidence of cirrhosis present
* Participants with hepatitis B core antibody positive must be on an antiviral agent to suppress hepatitis B throughout the study and be willing to continue therapy for at least one year after axicabtagene infusion
* Participants who are willing to continue ART during leukapheresis, manufacturing and infusion and post infusion of axicabtagene ciloleucel

Exclusion Criteria:

* Participants felt to have a high prospect of clinically benefiting from autologous transplantation
* Participants with central nervous system (CNS)-only involvement by malignancy (note: participants with secondary CNS involvement are allowed on study
* Participants with a second prior or concurrent malignancy that, in the opinion of the investigator, has a natural history or treatment course that has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Treatment with alemtuzumab within 6 months before anticipated leukapheresis, or treatment with fludarabine or cladribine within 3 months before anticipated leukapheresis
* Participants with uncontrolled systemic fungal, bacterial, viral, or other infection despite appropriate antibiotics or other treatment at the time of enrollment
* Presence of acute or chronic graft-versus-host disease
* History of any one of the following cardiovascular conditions within the past 6 months: class III or IV heart failure as defined by the New York Heart Association, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease
* History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
* Pregnant or nursing women. NOTE: Women of reproductive potential must have a negative serum pregnancy test performed within 48 hours before starting conditioning chemotherapy. Pregnant women are excluded from this study because axicabtagene ciloleucel has not been studied in pregnant women. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with axicabtagene ciloleucel, breastfeeding should be discontinued if the mother is treated with axicabtagene ciloleucel. These potential risks may also apply to other agents used in this study
* Use of the following:

  * Therapeutic doses of corticosteroids (defined as > 20 mg/day prednisone or equivalent) within 7 days before leukapheresis or 72 hours before axicabtagene ciloleucel administration. Physiologic replacement, topical, and inhaled steroids are permitted
  * Chemotherapy given after leukapheresis to maintain disease control must be stopped >= 7 days before conditioning chemotherapy
  * Cytotoxic chemotherapeutic agents that are not considered lymphotoxic (see below) within 1 week before leukapheresis. Oral chemotherapeutic agents, including lenalidomide and ibrutinib, are allowed if at least 3 half-lives have elapsed prior to leukapheresis
  * Lymphotoxic chemotherapeutic agents (e.g., cyclophosphamide, ifosfamide, bendamustine) within 2 weeks before leukapheresis
  * Experimental agents received within 4 weeks before leukapheresis unless no response or disease progression is documented while on the experimental therapy and at least 3 half-lives have elapsed before leukapheresis
  * Immunosuppressive therapies within 4 weeks before leukapheresis and axicabtagene ciloleucel administration (e.g., calcineurin inhibitors, methotrexate, or other chemotherapeutics, mycophenolate, rapamycin, thalidomide, immunosuppressive antibodies such as anti-TNF, anti-IL6, or anti-IL6R)
  * Donor lymphocyte infusions (DLI) within 6 weeks before axicabtagene ciloleucel administration
  * Radiation within 1 week before leukapheresis. Subjects must have progressive disease in irradiated lesions or have additional non-irradiated, PET-positive lesions to be eligible. However, palliative radiation to a single lesion, if additional non-irradiated PET-positive lesions are present, is allowed up to 2 weeks before leukapheresis
  * Prior receipt of CAR T-cell therapy
* Participants with signs or symptoms indicative of active CNS involvement are excluded from the protocol, with the following exceptions: The following patients are included in the protocol:

  * Participants with previously treated CNS involvement by lymphoma or leukemia, who and have no neurologic symptoms and no evidence of active lymphoma or leukemia in the CNS by total spine and brain gadolinium enhanced magnetic resonance imaging (MRI) within 2 weeks before leukapheresis and no neurologic progression prior to axicabtagene ciloleucel (axi-cel) infusion
  * Participants with active CNS involvement and stable neurologic symptoms for at least 3 weeks before leukapheresis and without neurologic progression prior to axi-cel infusion. These patients should have assessment by a total spine and brain gadolinium enhanced MRI within 5 days before axi-cel infusion to document the extent of CNS disease prior to axi-cel infusion. Cerebrospinal fluid (CSF) sampling for cell count, cytology and cell markers by flow cytometry should also be included within 5 days of axi-cel infusion if previously positive
* Inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Participants are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, including if >= 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted. Use of anabolic steroids is permitted
* The participant has not recovered to baseline or CTCAE =< grade 1 from toxicity due to all prior therapies except =< grade 2 alopecia, neuropathy, and other non-clinically significant adverse events (AEs), provided that all other eligibility criteria are met
* Opportunistic infection within the last 3 months, with the exception of oropharyngeal candidiasis
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to axicabtagene ciloleucel or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness with potential to limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety of chimeric antigen receptor (CAR) T-cell therapy | Up to 2 years
  Safety defined as blood count recovery of neutrophils and platelets to grade 2 or less within 6 weeks of CAR-T cell administration; incidence of infections; and cytokine release syndrome as defined by the 2019 American Society for Transplantation and Cellular Therapy harmonized system. The incidence of toxicity will be summarized using frequency and percentage and presented by overall and for each CD4 cohort.
Feasibility of CAR-T Therapy | Up to 2 years
  Feasibility defined as ability of enrolled participants in each cohort to receive axicabtagene ciloleucel. Feasibility will be estimated as the proportion of participants who receive axicabtagene ciloleucel among all enrolled participants who undergo leukapheresis. A two-sided 95% exact confidence interval will also be reported together with the estimated proportion. Production failure will be defined as the number of episodes of "inability to collect sufficient T-cells and/or create products." It will be summarized using descriptive statistics.

SECONDARY OUTCOMES:
Complete response rate | Up to 2 years
  Will be estimated as the proportion of participants who achieve complete response as per Lugano criteria. A two-sided exact 95% confidence interval will be reported together with the estimated response rate.
Event-free survival (EFS) | From time from randomization to earliest date of disease progression, commencement of new lymphoma therapy, or death, assessed up to 2 years
  EFS is defined as the time from randomization to the earliest date of disease progression per Lugano, commencement of new lymphoma therapy, or death from any cause. The event of interest includes disease progression or treatment discontinuation for any reason. Patients who do not experience an event will be censored at the last time the patient is alive without disease progression or treatment discontinuation. The distribution of event-free survival will be presented using Kaplan-Meier survival curves. The event-free survival probability together with 95% confidence interval at specific time points will be estimated using Kaplan-Meier method.
Duration of response (DOR) | From time when response criteria are met to the documentation of relapse or progression, assessed up to 2 years
  DOR defined as time from when response criteria (completer response or partial response) are met to the documentation of relapse or progression. The event of interest includes relapse, progression or death from any cause. For patients who die without disease, response duration is censored at the time of death. For patients who have not progressed, response duration is censored at the last time at which progression was assessed. The analysis approach for response duration will be similar to what has been described for event-free survival.
CD4 and CD8 counts | Up to 2 years
  The difference in CD4 and CD8 counts between those who achieve complete response and those who do not will be tested for statistical significance using Wilcoxon rank sum test. The analysis will be done for both CD4 count-based cohorts separately.

OTHER OUTCOMES:
Relationship between immune-mediated response and clinical response and toxicity in human immundeficiency virus (HIV)-associated B-Cell Non-Hodgkin Lymphoma treated with axicabtagene ciloleucel | Up to 2 years
  The difference between cytokine profiles and those who achieve complete response and those who do not as per Lugano criteria will be tested for statistical significance using Wilcoxon rank sum test. The association between cytokine profile and cytokine release syndrome status (>= grade 3 vs < grade 3) as well as immune effector cell-associated neurotoxicity (>= grade 3 vs < grade 3) will be tested for statistical significance using Wilcoxon rank sum test.
Burden of HIV integration in the final CAR T-cell product versus the pheresis product through quantitative polymerase chain reaction | Up to 2 years
  Will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Ariela Noy, Principal Investigator — AIDS Malignancy Consortium
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio state University, Columbus, Ohio
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah